CLINICAL TRIAL: NCT01537835
Title: Bacterial Contamination of Healthcare Worker Uniforms: A Study of Antimicrobial Uniforms on Occupationally Acquired Bacterial Contamination: A Randomized Controlled Trial
Brief Title: Bacterial Contamination of Healthcare Worker Uniforms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Denver Health and Hospital Authority (Other)
Collaborators: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2-5-15504
Record Dates: First submitted 2012-02-17; First posted 2012-02-23 (Estimated); Results first posted 2015-02-23 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Bacterial Contamination of Healthcare Worker Uniforms
Keywords: healthcare; worker; uniforms; bacterial; contamination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard Scrubs (No Intervention): Participants will be randomized to one of three types of uniforms. This arm is the standard scrub arm. The participants will wear new standard scrubs.
- Antimicrobial Scrubs 1 (Experimental): Participants will be randomized to one of three types of uniforms. In this arm, the participants will wear one of two types of antimicrobial uniforms. These are commercially available and registered with the Environmental Protective Agency.
  Interventions: Other: Antimicrobial Scrubs
- Antimicrobial Scrubs 2 (Experimental): Participants will be randomized to one of three types of uniforms. In this arm, the participants will wear one of two types of antimicrobial uniforms. These are commercially available and registered with the Environmental Protective Agency.
  Interventions: Other: Antimicrobial Scrubs

INTERVENTIONS:
Other: Antimicrobial Scrubs — Participants will be randomized to one of three types of scrubs. There will be a control (standard scrubs without antimicrobial properties) and two scrubs with reported antimicrobial properties.
  Arms: Antimicrobial Scrubs 1; Antimicrobial Scrubs 2

SUMMARY:
Healthcare worker uniforms are frequently contaminated with bacteria known to cause infections in humans. These bacteria are acquired during the workday. A new technology of antimicrobial textiles have been developed and incorporated into the fabric of health care worker uniforms, reportedly with effectiveness rates of > 99% but there is little literature describing the effectiveness of Healthcare worker (HCW) uniforms with antimicrobial properties in the clinical setting. Because of the potential benefit that such uniforms could offer HCWs and patients alike, further investigation into whether these fabrics are effective is warranted.

Up to 140 physicians, nurses, and midlevel providers who work at Denver Health on the general internal medicine wards will be invited to participate in this study. Participants will be randomized to wear either uniforms (scrubs) that have antimicrobial properties or standard scrubs provided by the hospital. At the end of an 8-hour workday, three areas on each uniform and each subject's wrist area will be cultured to assess for total bacterial colonization as well as for various resistant bacteria such as methicillin-resistant Staphylococcus aureus (MRSA), vancomycin-resistant Enterococcus (VRE), and resistant gram-negative rods.

Primary Hypothesis: HCW uniforms with antimicrobial properties will have less bacterial contamination than standard uniforms (scrubs) at the end of an 8-hour workday.

Specific aim 1a. Demonstrate that antimicrobial uniforms will have less total bacterial contamination of sites swabbed compared to standard uniform after an 8-hour workday.

Specific aim 1b. Demonstrate that antimicrobial uniforms will have less antimicrobial-resistant bacterial contamination (specifically looking for MRSA, VRE, and resistant gram negatives) of sites swabbed compared to standard uniform after an 8-hour workday.

ELIGIBILITY:
Inclusion Criteria:

* Physicians, nurses, and midlevel providers who work at Denver Health on the general internal medicine wards;
* Provider must be available for cultures at the end of the day, provider must be on service at Denver
* Health for the duration of the study, provider must be willing to avoid wearing white coats

Exclusion Criteria:

* Refusal to participate
* Known to be pregnant

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2011-11; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marisha A Burden, MD, Principal Investigator — Denver Health and Housing Authority
Locations (1):
- Denver Health and Hospital Authority, Denver, Colorado, United States

REFERENCES:
- [Background] Burden M, Cervantes L, Weed D, Keniston A, Price CS, Albert RK. Newly cleaned physician uniforms and infrequently washed white coats have similar rates of bacterial contamination after an 8-hour workday: a randomized controlled trial. J Hosp Med. 2011 Apr;6(4):177-82. doi: 10.1002/jhm.864. Epub 2011 Feb 10. PMID 21312328
- [Derived] Burden M, Keniston A, Frank MG, Brown CA, Zoucha J, Cervantes L, Weed D, Boyle K, Price C, Albert RK. Bacterial contamination of healthcare workers' uniforms: a randomized controlled trial of antimicrobial scrubs. J Hosp Med. 2013 Jul;8(7):380-5. doi: 10.1002/jhm.2051. Epub 2013 Jun 12. PMID 23757125

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Scrubs | Antimicrobial Scrubs 1 | Antimicrobial Scrubs 2
Started | 37 | 37 | 35
Completed | 37 | 37 | 35
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Please note two participants in the standard scrub group and two participants in the antimicrobial scrub group A were excluded from analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Scrubs | Antimicrobial Scrubs 1 | Antimicrobial Scrubs 2 | Total
Number analyzed (Participants) | 35 | 35 | 35 | 105
Age, Customized [Number; unit: participants] — Age was not collected.
  participants
    Not Available | NA — Age was not collected | NA — Age was not collected | NA — Age was not collected | NA — Total not calculated because data are not available (NA) in one or more arms.
Sex/Gender, Customized [Number; unit: participants] — Gender was not collected.
  participants
    Not Available | NA — Gender was not collected | NA — Gender was not collected | NA — Gender was not collected | NA — Total not calculated because data are not available (NA) in one or more arms.
healthcare worker type [Number; unit: participants]
  attending physician | 5 | 3 | 3 | 11
  intern/resident | 17 | 16 | 18 | 51
  midlevels | 2 | 2 | 2 | 6
  nurse | 11 | 14 | 12 | 37
cared for colonized or infected patient [Number; unit: participants] | 16 | 20 | 19 | 55

OUTCOME MEASURES:

1. Primary Outcome: Total Bacterial Contamination of Healthcare Worker Uniform With Antimicrobial Properties Compared to Standard Healthcare Worker Uniform After an 8-hour Workday.
Description: Total bacterial colony count of samples obtained from the breast or lower front pocket, the sleeve cuff of the dominant hand and the pant leg at the mid-thigh of the dominant leg on all scrubs after an eight-hour workday.
Time Frame: 8 hours
Population: healthcare workers randomized to one of three types of uniform.
Measure: Median (Inter-Quartile Range); unit: colony formation units
Arm/Group | Standard Scrubs | Antimicrobial Scrubs 1 | Antimicrobial Scrubs 2
Number analyzed (Participants) | 35 | 35 | 35
colony formation units | 41 [20 to 70] | 65 [35 to 117] | 41 [22 to 99]
Statistical Analysis 1: Comparison: Standard Scrubs vs Antimicrobial Scrubs 1 vs Antimicrobial Scrubs 2; Test type: Superiority or Other; p = 0.17, Kruskal-Wallis — p-value is adjusted for multiple comparisons

2. Secondary Outcome: Assess for Methicillin Resistent Staphylococcus Aureus, Vancomycin Resistant Enterococci, and Gram-negative Bacterial Contamination on Healthcare Worker Uniform With Antimicrobial Properties Compared to Standard Healthcare Worker Uniform.
Description: Number of healthcare workers with methicillin-resistant Staphylococcus aureus (MRSA), vancomycin-resistant enterococci (VRE), and resistant gram-negative bacteria on the three scrub types, all obtained after the eight-hour workday.
Time Frame: 8 hours
Population: Healthcare workers randomized to one of three types of uniform
Measure: Number; unit: participants
Arm/Group | Standard Scrubs | Antimicrobial Scrubs 1 | Antimicrobial Scrubs 2
Number analyzed (Participants) | 35 | 35 | 35
participants | 0 | 1 | 2

ADVERSE EVENTS:
Arm/Group | Standard Scrubs | Antimicrobial Scrubs 1 | Antimicrobial Scrubs 2
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 0/35 | 0/35 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No